CLINICAL TRIAL: NCT06889428
Title: Prognostic Significance of Cardiac Magnetic Resonance Imaging Confirmed Infarct in MINOCA Patients from Sweden and Australia
Brief Title: Prognostic Significance of CMR-Confirmed Infarct in MINOCA Patients from Sweden and Australia
Acronym: SWEET
Status: Completed | Type: Observational
Sponsor: University of Adelaide (Other)
Collaborators: Uppsala University (Other)
Responsible Party: Principal Investigator, Sivabaskari Pasupathy, Principal Investigator (Research Fellow), University of Adelaide
Other Study IDs: HREC/15/TQEH/252 - SWEET
Record Dates: First submitted 2025-03-10; First posted 2025-03-21 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: MINOCA
Keywords: cardiac magnetic resonance imaging; prognosis; Myocarditis
MeSH Terms: conditions — MINOCA; Myocarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Suspected MINOCA with CMR: Patients who have undergone a CMR procedure as part of their care at the time of acute presentation with MI.
  Interventions: Diagnostic Test: CMR
- Suspected MINOCA without CMR: Patients who did not undergo a CMR procedure as part of their care at the time of acute presentation with MI.
- Patients with confirmed MINOCA: Suspected MINOCA patients who have received a diagnosis of MI following CMR
  Interventions: Diagnostic Test: CMR
- Patients with other CMR diagnosis: Suspected MINOCA patients who did not receive a diagnosis of MI following CMR

INTERVENTIONS:
Diagnostic Test: CMR — No CMR
  Other Names: Cardiac magnetic resonance imaging; Cardiac MRI
  Groups: Patients with confirmed MINOCA; Suspected MINOCA with CMR

SUMMARY:
Myocardial Infarction (MI) with Non-Obstructive Coronary Arteries (MINOCA), occurring in 6-8% of MIs, refers to patients who experience a heart attack without obstructive coronary artery disease (CAD) or significant atherosclerosis. One of the challenges inherent to MINOCA lies in its propensity to mimic non-coronary-related pathologies, such as myocarditis or takotsubo. Thus, Cardiac Magnetic Resonance (MRI) imaging has been recommended as the central diagnostic tool for confirming MINOCA diagnosis while excluding the others. However, the resource-intensive nature of MRI, combined with its limited availability in hospitals, poses barriers to patient access and limits research activities that could produce significant impact. Therefore, this project's aim is to curate the largest dataset of suspected MINOCA patients with MRI, via a collaboration between Sweden's nationwide registry and South Australia's state-wide registry, to answer the following key questions: (i) What is prognosis of MINOCA, as confirmed by MRI? (ii) What are the characteristics and prognosis of patients who had MRI compared to those who did not? (iii) What clinical parameters are associated with MINOCA on MRI?

This project will utilize DataSHIELD, an innovative platform that enables pooled statistical analysis of sensitive data without compromising individual-level privacy. This multicentre, comprehensive study will have a major impact on contemporary practice. It will be able to provide the significance of MINOCA diagnosis (myocardial scar on MRI), alongside identifying clinical factors associated with its occurrence and its correlation with long-term outcomes.

This is crucial for informing clinical guidelines, policy decisions around reimbursement for MRI, and developing effective clinical trials to enhance the management of MRI-confirmed MINOCA patients

ELIGIBILITY:
Inclusion Criteria:

1. Discharge diagnosis of MINOCA - acute presentation with (a) universal criteria for acute MI (b) non-obstructive coronaries on angiography.
2. Cardiac MRI - at least within 3 months of acute presentation

Exclusion Criteria:

1. Patients without satisfactory images on cardiac MRI
2. Follow-up data not available (ie international visitors).
3. Suspicion of an alternative cause for presentation (such as sepsis, pulmonary embolus, primary cardiac arrhythmia or trauma) which would not be consistent with the label of MINOCA.
4. Clinically evident non-ischemic diagnoses - myocarditis, Takotsubo, other cardiomyopathies prior to CMR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The data will extracted from CADOSA and SWEDEHEART registries for the purpose of this study.
  * CADOSA (Australia): The Coronary Angiogram Database Of South Australia registry is highly robust, collecting detailed and comprehensive information on patients undergoing coronary angiogram procedure in South Australia. It includes patient features, comorbidities, chest pain and ECG characteristics, coronay angiogram details, admission/discharge medications etc. Data is collected directly from patients and medical records in real-time by trained collectors, ensuring data quality and reliability.
  * SWEDEHEART (Sweden): The Swedish Web-system for Enhancement and Development of Evidence-based care in Heart disease Evaluated According to Recommended Therapies (SWEDEHEART) registry is a comprehensive and nationwide registry in Sweden that focuses on the management and treatment of patients with cardiovascular diseases.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Experiencing Major Adverse Cardiovascular Events (MACE) | 36 Months
  The proportion of participants experiencing the first occurrence of MACE, defined as all-cause mortality, cardiac mortality, myocardial infarction, unstable angina, heart failure hospitalization, or stroke following MINOCA.

SECONDARY OUTCOMES:
Percentage of Participants with All-Cause Mortality | 36 Months
  Proportion of participants who experience death from any cause following MINOCA.
Percentage of Participants with Cardiac Mortality | 36 Months
  Proportion of participants who experience death due to a cardiac cause following MINOCA
Percentage of Participants with Myocardial Infarction (Re-Infarction) | 36 Months
  Proportion of participants who are re-admitted for myocardial infarction following MINOCA
Percentage of Participants with Hospital admission for Unstable Angina | 36 Months
  Proportion of participants who are admitted for unstable angina following MINOCA.
Percentage of Participants Hospitalized for Heart Failure | 36 Months
  The proportion of participants who require hospitalization due to heart failure following MINOCA
Percentage of Participants Experiencing a Stroke | 36 Months
  The proportion of participants who experience a stroke following MINOCA
Percentage of Participants with All-Cause Mortality | 12 Months
  Proportion of participants who experience death from any cause following MINOCA.
Percentage of Participants with Cardiac Mortality | 12 Months
  Proportion of participants who experience death due to a cardiac cause following MINOCA
Percentage of Participants with Myocardial Infarction (Re-Infarction) | 12 Months
  Proportion of participants who are re-admitted for myocardial infarction following MINOCA
Percentage of Participants with Hospital admission for Unstable Angina | 12 Months
  Proportion of participants who are admitted for unstable angina following MINOCA.
Percentage of Participants Hospitalized for Heart Failure | 12 Months
  The proportion of participants who require hospitalization due to heart failure following MINOCA
Percentage of Participants Experiencing a Stroke | 12 Months
  The proportion of participants who experience a stroke following MINOCA
Percentage of Participants Presenting to the Emergency Department with Chest Pain | 36 Months
  The proportion of participants who present to the emergency department with chest pain, expressed as a percentage of the total study population.
Percentage of Participants Presenting to the Emergency Department with Chest Pain | 12 Months
  The proportion of participants who present to the emergency department with chest pain, expressed as a percentage of the total study population.
Percentage of Participants with Late Gadolinium Enhancement (LGE) Features on CMR Following suspected MINOCA | From CMR performed within 3 months from acute presentation
  The proportion of participants with detectable LGE on cardiac magnetic resonance (CMR) , indicating myocardial fibrosis or necrosis.
Percentage of Participants with Abnormal Tissue Characteristics on CMR in Suspected MINOCA | From CMR performed within 3 months from acute presentation
  The proportion of participants with suspected MINOCA who exhibit abnormal myocardial tissue characteristics on CMR, including myocardial edema,
Percentage of Participants with Evidence of Myocarditis on CMR in Suspected MINOCA | From CMR performed within 3 months from acute presentation
  The proportion of participants with suspected MINOCA who have CMR findings consistent with myocarditis (e.g., myocardial edema, LGE patterns suggestive of inflammation).
Percentage of Participants with Evidence of Takotsubo Syndrome on CMR in Suspected MINOCA | From CMR performed within 3 months from acute presentation
  The proportion of participants with suspected MINOCA who demonstrate CMR findings consistent with Takotsubo syndrome (e.g., apical ballooning, absence of LGE).
Percentage of Participants with Normal CMR Findings in Suspected MINOCA | From CMR performed within 3 months from acute presentation
  The proportion of participants with suspected MINOCA who have no significant abnormalities on CMR, indicating no structural or ischemic myocardial injury.

CONTACTS AND LOCATIONS:
Overall Officials: John Beltrame, PhD, Principal Investigator — University of Adelaide; Bertil Lindahl, Principal Investigator — Uppsala University; Sivabaskari Pasupathy, PhD, Principal Investigator — University of Adelaide
Locations (1):
- University of Adelaide, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No
For privacy reasons, the IPD will not be shared between countries